CLINICAL TRIAL: NCT06569043
Title: Appetite Responses to Breakfast Bar Product: a Randomized Controlled Trial
Brief Title: Appetite Responses to Breakfast Bar Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Mills (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 597
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Satisfaction, Consumer
MeSH Terms: conditions — Consumer Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Breakfast Bar (Experimental): Packaged breakfast bar available in retail stores
  Interventions: Other: Breakfast Bar
- Control (No Intervention): No intervention (i.e., no food provided)

INTERVENTIONS:
Other: Breakfast Bar — Packaged breakfast bar product available in retail stores
  Arms: Breakfast Bar

SUMMARY:
The purpose of this clinical trial is to investigate appetite responses to 2 cereal products in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-70 years
* Habitual snack bar consumers (at least several times per month)
* Body mass index 18.5-29.9 kg/m2 (based on self-reported weight and height)
* Understand and willing to follow the study procedures
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial
* Willing to abstain from strenuous exercise, consuming alcoholic drinks 24 hours before the test day
* Willing to provide informed consent to participate in the study

Exclusion Criteria:

* Pregnant or lactating women, or women who are planning to become pregnant during the study
* Known food allergies, sensitivities, or intolerance to any food or food ingredients
* Participating in another clinical trial for food, investigational drug, nutritional supplement, or lifestyle modification
* Taking medications that affect appetite, metabolism or blood pressure
* Presence of acute diseases or infection
* Presence or history of chronic diseases
* Diagnosed with an eating disorder
* Restraint eaters as determined by a score >4 from the Dutch Eating Behavior Questionnaire
* Lost or gained 5 or more pounds in the past 3-months
* On a weight loss diet or undergoing intermittent fasting
* COVID-19 infection within the past 3 months
* Subjects who do not eat bar products

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-10-20 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale for Hunger 0-240 minutes | 240 minutes
  Visual Analogue Scale for "how hungry are you right now?" is scored from 0-100 millimeters (mm), whereby a higher mm indicates more hunger. Comparing change from 0 minutes (baseline) to 240 minutes, whereby a lower mm change from baseline indicates a better outcome.
Visual Analogue Scale for Fullness 0-240 minutes | 240 minutes
  Visual Analogue Scale for "how full are you right now?" is scored from 0-100 millimeters (mm), whereby a higher mm indicates more fullness. Comparing change from 0 minutes (baseline) to 240 minutes, whereby a higher mm change from baseline indicates a better outcome.
Visual Analogue Scale for Satiation 0-240 minutes | 240 minutes
  Visual Analogue Scale for "how satiated are you right now?" is scored from 0-100 millimeters (mm), whereby a higher mm indicates more satiation. Comparing change from 0 minutes (baseline) to 240 minutes, whereby a higher mm change from baseline indicates a better outcome.
Visual Analogue Scale for Desire to Eat 0-240 minutes | 240 minutes
  Visual Analogue Scale for "how strong is your desire to eat right now?" is scored from 0-100 millimeters (mm), whereby a higher mm indicates more desire to eat. Comparing change from 0 minutes (baseline) to 240 minutes, whereby a lower mm change from baseline indicates a better outcome.
Visual Analogue Scale for Prospective Consumption 0-240 minutes | 240 minutes
  Visual Analogue Scale for "how much do you think you can eat right now?" is scored from 0-100 millimeters (mm), whereby a higher mm indicates more prospective consumption. Comparing change from 0 minutes (baseline) to 240 minutes, whereby a lower mm change from baseline indicates a better outcome.
Visual Analogue Scale for Satisfaction 0-240 minutes | 240 minutes
  Visual Analogue Scale for "how satisfied are you right now?" is scored from 0-100 millimeters (mm), whereby a higher mm indicates more satisfaction. Comparing change from 0 minutes (baseline) to 240 minutes, whereby a higher mm change from baseline indicates a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Remote, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No